CLINICAL TRIAL: NCT04952064
Title: Ganglioside GM1 in Acute Ischemic Stroke: a Prospective, Randomized, Blinded Assessment of Endpoints, and Multicenter Exploratory Study
Brief Title: An Exploratory Study of Ganglioside GM1 in Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Collaborators: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y（2021）052
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Stroke, Ischemic
Keywords: monosialoganglioside GM1; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 200 mg group (Experimental): Monosialoganglioside GM1, 200 mg/day, for 12-14 days
  Interventions: Drug: Monosialoganglioside GM1
- 400 mg group (Experimental): Monosialoganglioside GM1, 400 mg/day, for 12-14 days
  Interventions: Drug: Monosialoganglioside GM1

INTERVENTIONS:
Drug: Monosialoganglioside GM1 — Monosialoganglioside GM1 diluted with 0.9% normal saline 100ml, iv, daily for 12-14 days
  Other Names: GM1

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of higher doses of monosialoganglioside GM1 injection in the treatment of patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-80 years old；
* 2. Patients with anterior circulation cerebral infarction;
* 3. first stroke onset or past stroke without obvious neurological deficit (mRS score≤1)；
* 4. Within 24 hours of onset；
* 5. 5 ≤NIHSS score ≤ 20；
* 6. Signed informed consent.

Exclusion Criteria:

* 1. Patients with hereditary abnormal glucose and lipid metabolism (gangliosidosis, such as Tay-Sachs disease and retinal degeneration);
* 2. Hemorrhagic stroke;
* 3. Disturbance of consciousness (NIHSS1a≥1)，or cerebral arteritis, brain tumor, brain trauma, intracranial infectious diseases;
* 4. Planed endovascular treatment;
* 5. Uncontrolled hypertension: systolic pressure ≥200 mmHg or diastolic pressure ≥110 mmHg;
* 6. Bleeding tendency (except for thrombolysis) or severe bleeding within 3 months;
* 7. Patients with malignant tumor or serious diseases;
* 8. Along with epilepsy, arthritis and other disease, which have effect on neurological assessment;
* 9. History of autoimmune diseases, spinal trauma, various demyelinating diseases, including acute inflammatory demyelinating polyneuropathy (Guillain Barre syndrome);
* 10. Unable or unwilling to cooperate due to mental diseases;
* 11. Abnormal liver and renal function: ALT, AST > 2 times of the upper limit of normal value, or Cr > 1.5 times of the upper limit of normal value；
* 12. Hypersensitivity to monosialoganglioside and excipients of test drug;
* 13. History of drug abuse；
* 14. Pregnant or lactating women, pregnant plan or unwilling to use effective contraception during the trial period;
* 15. Participating in other clinical trials within 3 months;
* 16. Other conditions which are unsuitable for this trial assessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-2 | 90 days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome

SECONDARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-1 | 90 days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome
changes in National Institute of Health stroke scale | 7 days and 14 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
changes in Barthel index (BI) scale | 30 days and 90 days
  the minimum and maximum values of BI are 0 and 100, respectively; higher BI mean a good outcome

OTHER OUTCOMES:
changes in some serum biomarkers | 7 days and 14 days
  serum biomarkers included SOD，BDNF，NGF，CRP，TNF-α，IL-6，IL-1β，VEGF，NO，MMP
The change of infarct volume | 3 days
  The change of infarct volume showed by MRI compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chen Huisheng, Doctor, Study Chair — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, Liaoning, China